CLINICAL TRIAL: NCT00438971
Title: The Efficacy and Tolerability of Duloxetine for the Treatment of Panic Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Mark H. Pollack, The Efficacy and Tolerability of Duloxetine for the Treatment of Panic Disorder, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-P-000263
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Results first posted 2013-12-19 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-03

CONDITIONS: Panic Disorder
Keywords: Panic Disorder; Anxiety Disorder; Duloxetine
MeSH Terms: conditions — Panic Disorder; Anxiety Disorders | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Duloxetine (Experimental)
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — Treatment will be initiated at 30mg/day in the first week (week 0), and then increased to 60mg/day at week 1, with the option to increase to 90mg at week 4, and 120mg at week 6.
  Other Names: Cymbalta

SUMMARY:
The purpose of this study is to determine whether duloxetine is effective in the treatment of panic disorder.

DETAILED DESCRIPTION:
Panic Disorder is relatively common, with a lifetime prevalence of 3.5 % (Kessler, et al 1994) and characterized by a typically chronic course (Marzol & Pollack, 2000). Affected individuals tend to be high utilizers of general health care services, frequently receiving extensive and unrevealing medical work-ups (Katon, 1997); while the panic disorder itself often goes unrecognized (Sartorious, et al 1993). Panic disorder has a significant negative impact on work, family, and social life (Rubin, et al 2000), and is associated with increased rates of negative life events and diminished overall quality of life (Cramer, et al 2005). Research indicates that the quality of life and well-being of patients with panic disorder is similarly or more impaired than that of patients with serious medical illnesses, such as type II diabetes (Rubin, et al 2000).

Treatment of panic disorder is focused on the reduction of panic attacks, avoidance behavior, and anticipatory anxiety, as well as the resolution of comorbid conditions. The overarching goal of panic disorder treatment is reduction in symptoms to allow improvement in overall quality of life (Pollack, 2005).

Duloxetine is a serotonin-norepinephrine reuptake inhibitor (SNRI) that has greater initial noradrenergic effects than venlafaxine (Goldstein, et al 2004). Recent data from a placebo controlled fixed dose study, suggested that venlafaxine at 225 mg/d (a dose at which noradrenergic effects are likely to be relevant), was more efficacious on a number of measures of panic disorder than the SSRI, paroxetine (Pollack, et al 2003). This data, combined with our clinical experience with duloxetine to date, support the assertion that duloxetine is likely to prove an effective agent for panic disorder.

Thus, we propose to perform the first systematic examination of the efficacy of duloxetine for panic disorder in a study in which 15 patients with panic disorder will receive duloxetine flexibly dosed from 30 to 120 mg/d in open treatment for 8 weeks. Information learned in this study will help guide treatment selection for panic disorder by providing initial open efficacy data for duloxetine in panic disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients, age 18-75.
* Diagnosis of Panic Disorder with or without Agoraphobia by DSM-IV criteria
* MGH Panic Clinical Global Impression of Severity score Score equal to or greater than 4
* Patients with current major depressive disorder will be allowed if the panic disorder is primary (as determined on interview by clinician and patient), and the baseline MADRS score is less than or equal to 20
* Willingness and ability to comply with the requirements of the study protocol.

Exclusion Criteria:

* Pregnant or lactating women or others not using acceptable means of birth control (e.g., IUD, oral contraceptives, barrier devices, condoms and foam, implanted progesterone rods stabilized for at least 3 months).
* Patients with current or history of posttraumatic stress disorder, obsessive compulsive disorder, bipolar disorder, schizophrenia or other psychotic conditions.
* Patients on other psychoactive medication, including MAOIs, and those with the potential need to use an MAOI during the study or within 5 day of discontinuation of study drug will be excluded. Participants must have discontinued MAOI use at least 14 days prior study baseline. Patients must discontinue regular benzodiazepine or other non-MAOI antidepressant therapy at least one week (5 weeks for fluoxetine) prior to baseline. Concomitant beta-blockers are proscribed unless prescribed for a medical indication (e.g., hypertension, at a stable daily dose for > 1 month).
* Patients with a history of alcohol or substance abuse or dependence within the last twelve months, significant alcohol dependence, or a positive toxicology screen consistent with abuse at baseline.
* Patients with significant or unstable neurological or medical disorders or instability for which hospitalization may be likely within the next year. In particular, patients with end-stage renal disease (requiring dialysis) or severe renal impairment, or hepatic insufficiency (defined as twice normal on LFTs as follows: SGPT >110 u/L or SGOT >80 u/L) will be excluded.
* Patients with uncontrolled narrow-angle glaucoma will be excluded.
* Seizure disorders with the exception of a history of febrile seizures if they occurred during childhood, were isolated, and did not recur in adulthood.
* Severe personality disorders likely to interfere with study participation.
* Ongoing psychotherapy directed toward the treatment of the panic disorder or agoraphobia. Prohibited psychotherapy includes cognitive behavioral therapy or psychodynamic therapy that focuses on exploring specific, dynamic causes of the panic or phobic symptoms and provides skills for their management, or any of the active ingredients of these psychotherapies. General supportive individual, couples, or family therapy greater than 2 months duration is acceptable.
* History of hypersensitivity or prior non-response or intolerance of duloxetine.
* Patients who have failed 4 or more medication trials of at least 4 weeks at adequate dose (e.g. paroxetine 20mg or equivalent). Treatment failure is here defined as clinician judgment based on assessment of patient history of prior treatment of minimal or no reduction in panic attacks, anticipatory anxiety or avoidance during a specific, medication trial.
* Patients with significant suicidal ideation (MADRS item 10 score > 3) or who have enacted suicidal behaviors within 6 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Pollack, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- The Center for Anxiety and Traumatic Stress Disorders at Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Kessler RC, McGonagle KA, Zhao S, Nelson CB, Hughes M, Eshleman S, Wittchen HU, Kendler KS. Lifetime and 12-month prevalence of DSM-III-R psychiatric disorders in the United States. Results from the National Comorbidity Survey. Arch Gen Psychiatry. 1994 Jan;51(1):8-19. doi: 10.1001/archpsyc.1994.03950010008002. PMID 8279933
- [Background] Marzol PC, Pollack MH. New developments in panic disorder. Curr Psychiatry Rep. 2000 Aug;2(4):353-7. doi: 10.1007/s11920-000-0081-8. PMID 11122981
- [Background] Katon W, Hart R, Montano B. The effect of panic disorder in the managed care setting. Manag Care Interface. 1997 Nov;10(11):88-94, 98. PMID 10174760
- [Background] Sartorius N, Ustun TB, Costa e Silva JA, Goldberg D, Lecrubier Y, Ormel J, Von Korff M, Wittchen HU. An international study of psychological problems in primary care. Preliminary report from the World Health Organization Collaborative Project on 'Psychological Problems in General Health Care'. Arch Gen Psychiatry. 1993 Oct;50(10):819-24. doi: 10.1001/archpsyc.1993.01820220075008. PMID 8215805
- [Background] Rubin HC, Rapaport MH, Levine B, Gladsjo JK, Rabin A, Auerbach M, Judd LL, Kaplan R. Quality of well being in panic disorder: the assessment of psychiatric and general disability. J Affect Disord. 2000 Jan-Mar;57(1-3):217-21. doi: 10.1016/s0165-0327(99)00030-0. PMID 10708834
- [Background] Cramer V, Torgersen S, Kringlen E. Quality of life and anxiety disorders: a population study. J Nerv Ment Dis. 2005 Mar;193(3):196-202. doi: 10.1097/01.nmd.0000154836.22687.13. PMID 15729110
- [Background] Pollack MH. The pharmacotherapy of panic disorder. J Clin Psychiatry. 2005;66 Suppl 4:23-7. PMID 15842184
- [Background] Pollack MH, Meoni P, Otto MW, Simon N, Hackett D. Predictors of outcome following venlafaxine extended-release treatment of DSM-IV generalized anxiety disorder: a pooled analysis of short- and long-term studies. J Clin Psychopharmacol. 2003 Jun;23(3):250-9. doi: 10.1097/01.jcp.0000084025.22282.84. PMID 12826987
- [Background] Goldstein DJ, Lu Y, Detke MJ, Wiltse C, Mallinckrodt C, Demitrack MA. Duloxetine in the treatment of depression: a double-blind placebo-controlled comparison with paroxetine. J Clin Psychopharmacol. 2004 Aug;24(4):389-99. doi: 10.1097/01.jcp.0000132448.65972.d9. PMID 15232330
- [Result] Simon NM, Kaufman RE, Hoge EA, Worthington JJ, Herlands NN, Owens ME, Pollack MH. Open-label support for duloxetine for the treatment of panic disorder. CNS Neurosci Ther. 2009 Winter;15(1):19-23. doi: 10.1111/j.1755-5949.2008.00076.x. PMID 19228176

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatients 18-75 years of age with a current DSM-IV diagnosis of panic disorder with or without agoraphobia were recruited through hospital and media advertisement between August 2006 and April 2008.
Pre-assignment Details: Subjects were required to be free of all psychiatric medications except for benzodiazepines initiated at least 2 weeks prior to study initiation and with the dose held stable during the trial. Of the 17 individuals initially enrolled, 2 completed the screening procedure but did not initiate pharmacotherapy and are not included in analyses.
Groups:
- Duloxetine: Duloxetine was initiated at 30 mg/day at the baseline visit, flexibly increased to 60 mg/day after 1 week, then flexibly titrated up to a maximum of 120 mg/day over the next 4 weeks based on response and tolerability with a minimum dose of 60 mg by week 4 required in order for the patient to remain in the study.
Period: Overall Study
Arm/Group | Duloxetine
Started | 17
Completed | 15
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Duloxetine
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 15
Panic Disorder Severity Scale (PDSS) - Primary Outcome [Mean (Standard Deviation); unit: units on a scale] | 14.2 (4.28)
Clinical Global Impression of Severity scale (CGI-S) [Mean (Standard Deviation); unit: units on a scale] | 4.80 (0.67)
Panic Attack Scale (PAS) [Mean (Standard Deviation); unit: units on a scale] | 3.90 (2.38)

OUTCOME MEASURES:

1. Primary Outcome: Panic Disorder Severity Scale (PDSS)
Description: The PDSS contains seven items assessing multiple dimensions of panic disorder severity, including (a) frequency of panic attacks, (b) distress during panic attacks, (c) anticipatory anxiety, (d) agoraphobic fear and avoidance, (e) interoceptive fear and avoidance, (f) impairment of work functioning, and (g) impairment of social functioning. The PDSS ranges from 0 to 28, with higher ratings reflecting greater degrees of symptom severity.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 15
units on a scale | 9.13 (5.26)

2. Secondary Outcome: Clinical Global Impression of Severity Scale (CGI-S)
Description: The CGI-S is a clinician-rated instrument used to assess global severity of symptoms. The CGI-S ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill). Remission was defined strictly as a CGI-S score of 1 or 2 (not at all ill or borderline ill) and zero panic attacks at endpoint.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 15
units on a scale | 3.47 (1.3)

3. Secondary Outcome: Panic Attack Scale (PAS)
Description: The PAS is a measure that assesses participants' total number of panic attacks (situational and unexpected with full and limited symptoms), as well as anticipatory anxiety, since last visit. There is no total score.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 15
units on a scale | 0.90 (1.44)

4. Other Pre Specified Outcome: Montgomery Asberg Depression Rating Scale (MADRS)
Description: The MADRS is a 10-item clinician rating of depressive symptoms. Scores range from 0 to 60, with higher scores reflecting greater symptom severity.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 15
units on a scale | 9.07 (6.68)

5. Other Pre Specified Outcome: Beck Anxiety Inventory (BAI)
Description: The BAI is a 21-item self-report measure of anxiety with a focus on somatic symptoms. Total scores range from 0 to 63, with higher scores reflecting greater symptom severity.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 15
units on a scale | 14.7 (13.7)

6. Other Pre Specified Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q)
Description: The Q-LES-Q is a self-report measure of the degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning. Only the first 14 items are included in scoring, which ranges from 14 to 70, with higher scores reflecting greater enjoyment and satisfaction. The last two items are not included in the total score but are standalone items.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 15
units on a scale | 49.3 (12.8)

7. Other Pre Specified Outcome: Sheehan Disability Scale (SDS)
Description: The SDS is a 3-item measure with each item rated on a 10-point scale. The SDS measures the extent to which work/school, social life, and home life or family responsibilities are impaired by symptoms. Total scores range from 0 to 30, with higher scores reflecting greater impairment.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 15
units on a scale | 9.40 (8.61)

8. Other Pre Specified Outcome: Longitudinal Interval Follow-up Evaluation Range of Impaired Functioning Tool (LIFE-RIFT)
Description: The LIFE-RIFT is a brief measure of psychosocial functioning in work, interpersonal relations, satisfaction, and recreation. Scores on the LIFE-RIFT can range from 4, indicating very good functioning (no impairment) in all of the 4 component areas, to 20, indicating very poor functioning (severe impairment) in all of the 4 areas.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 15
units on a scale | 9.33 (3.63)

ADVERSE EVENTS:
Arm/Group | Duloxetine
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=15)
Increased Anxiety Leading to Hospitalization (General disorders) | 1 (1) — Patient presented to the Emergency Department with increased panic attacks and anxiety after he called EMS for another student with a suspected injury. This situational increase in anxiety was not likely to be associated with study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duloxetine (N=15)
Appetite Decrease (General disorders) | 1
Appetite Increase (General disorders) | 1
Constipation (General disorders) | 2
Dry Mouth (General disorders) | 2
Dyspepsia (General disorders) | 1
Nausea (General disorders) | 3
Weight Gain (General disorders) | 1
Blurred Vision (General disorders) | 1
Headache (General disorders) | 2
Jitteriness (General disorders) | 2
Anxiety (General disorders) | 1
Sexual Dysfunction (General disorders) | 3
Urinary Hesitation (General disorders) | 2
Insomnia (General disorders) | 2
Sedation (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No